CLINICAL TRIAL: NCT03713320
Title: SOLAR: A Phase 2, Randomized, Open-label, Parallel-group, Active Comparator, Multi-center Study to Investigate the Efficacy and Safety of Cobomarsen (MRG-106) in Subjects With Cutaneous T-Cell Lymphoma (CTCL), Mycosis Fungoides (MF) Subtype
Brief Title: SOLAR: Efficacy and Safety of Cobomarsen (MRG-106) vs. Active Comparator in Subjects With Mycosis Fungoides
Acronym: SOLAR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early for business reasons, and not due to concerns regarding safety or lack of efficacy.
Sponsor: miRagen Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRG106-11-201; 2018-000727-13 (EudraCT Number)
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Results first posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Cutaneous T-Cell Lymphoma/Mycosis Fungoides
Keywords: SOLAR; Cutaneous T-cell Lymphoma; CTCL; Mycosis Fungoides; Lymphoma; Lymphoma, T-cell; Lymphoma, T-cell, cutaneous; Lymphoma, Non-Hodgkin; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Neoplasms; MicroRNAs; Vorinostat; Histone Deacetylase Inhibitors
MeSH Terms: conditions — Mycosis Fungoides; Lymphoma, T-Cell, Cutaneous; Lymphoma; Lymphoma, T-Cell; Lymphoma, Non-Hodgkin; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Neoplasms | interventions — cobomarsen; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cobomarsen (Experimental): Cobomarsen will be administered by intravenous 2-hour infusion at a dose of 282 mg on Days 1, 3, 5, 8, and weekly thereafter
  Interventions: Drug: Cobomarsen
- Vorinostat (Active Comparator): Vorinostat will be administered orally at a dose of 400 mg (four 100-mg capsules) once daily with food, at approximately the same time each day.
  Interventions: Drug: Vorinostat

INTERVENTIONS:
Drug: Cobomarsen — At least weekly doses of cobomarsen (282 mg) throughout study treatment period
  Other Names: MRG-106
  Arms: Cobomarsen
Drug: Vorinostat — Daily doses of vorinostat throughout study treatment period
  Arms: Vorinostat

SUMMARY:
The main objective of this clinical trial is to study the efficacy and safety of cobomarsen (also known as MRG-106) for the treatment of cutaneous T-cell lymphoma (CTCL), mycosis fungoides (MF) subtype. Cobomarsen is designed to inhibit the activity of a molecule called miR-155 that may be important to the growth and survival of MF cancer cells. The study will compare the effects of cobomarsen to vorinostat, a drug that has been approved for the treatment of CTCL in the United States and several other countries.

Participants in the clinical trial will be randomly assigned to receive either weekly doses of cobomarsen by injection into a vein or daily oral doses of vorinostat. Participants will continue on their assigned treatment as long as there is no evidence of progression of their cancer. The effects of treatment will be measured based on changes in skin lesion severity, as well as the length of time that the subject's disease remains stable or improved, without evidence of disease progression. The safety and tolerability of cobomarsen will be assessed based on the frequency and severity of observed side effects.

Participants assigned to receive vorinostat who experience progression of their disease during their participation in this study may have the option to be treated with cobomarsen in an open-label, crossover arm of the same study if they meet the entry criteria for that part of the study.

DETAILED DESCRIPTION:
Study Design:

Subjects will be randomly assigned in a 1:1 ratio to receive either cobomarsen or vorinostat. Approximately 126 subjects (63 per arm) are expected to be enrolled. Cobomarsen will be administered in the clinic by 2-hr intravenous infusion on Days 1, 3, 5 and 8, and weekly thereafter. Vorinostat will be dispensed to study subjects and taken as a daily oral dose according to the manufacturer's labeled dosing instructions. Treatment will continue until the subject becomes intolerant, develops clinically significant side effects, progresses, or the trial is terminated. An interim analysis will be conducted after approximately 40 subjects have been followed for a minimum of approximately 6 months. Enrollment will be suspended until the completion of the interim analysis.

ELIGIBILITY:
Key Inclusion Criteria:

* Biopsy-proven CTCL, MF subtype
* Clinical stage IB, II, or III, with staging based on screening assessments
* Minimum mSWAT score of 10 at screening
* Receipt of at least one prior therapy for CTCL

Key Exclusion Criteria:

* Previous enrollment in a cobomarsen study
* Prior therapy with vorinostat or other HDAC inhibitors, or contraindication to an HDAC inhibitor
* Sézary syndrome or mycosis fungoides with B2 involvement, defined as documented history of B2 and/or B2 staging at screening
* Evidence of large cell transformation
* Lymph node involvement at screening, unless radiologically or histologically confirmed to be nonmalignant
* Visceral involvement related to MF at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2020-10-12 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana M. Escolar, MD, FAAN, Study Director — miRagen Therapeutics, Inc.
Locations (43):
- United States (20):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic, Phoenix, Arizona
  - City of Hope, Duarte, California
  - UCLA, Los Angeles, California
  - Chao Family Comprehensive Cancer Center at University of California, Irvine, Orange, California
  - Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - Mayo Clinic, Jacksonville, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Rochester Skin Lymphoma Medical Group, Fairport, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - University of Washington, Seattle, Washington
- Australia (3):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Linear Clinical Research, Nedlands
- University Clinic UZ Leuven, Leuven, Belgium
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - Jewish General Hospital, Montreal, Quebec
- France (5):
  - Hôpital Saint André, CHU de Bordeaux, Bordeaux
  - Hôpital Saint-Louis, Paris
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Hôpital Robert Dubré, CHU de Reims, Reims
  - Centre Hospitalier Universitaire de Rouen, Rouen
- Italy (3):
  - Policlinico S. Orsola-Malpighi, Bologna
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - AOU Citta dell Salute e della Scienza di Torino, Torino
- Spain (5):
  - Vall d'Hebron Institute of Oncology, Barcelona
  - Fundación Jiménez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Consorcio Hospital General Universitario Valencia, Valencia
- United Kingdom (4):
  - University Hospitals of Birmingham NHS Foundation Trust, Queen Elizabeth Hospital, Birmingham
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Guy's and St. Thomas' NHS Foundation Trust, Cancer Center, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ganguly K, Kishore U, Madan T. Interplay between C-type lectin receptors and microRNAs in cellular homeostasis and immune response. FEBS J. 2021 Jul;288(14):4210-4229. doi: 10.1111/febs.15603. Epub 2020 Nov 7. PMID 33085815
- [Derived] Valipour A, Jager M, Wu P, Schmitt J, Bunch C, Weberschock T. Interventions for mycosis fungoides. Cochrane Database Syst Rev. 2020 Jul 7;7(7):CD008946. doi: 10.1002/14651858.CD008946.pub3. PMID 32632956

RESULTS

PARTICIPANT FLOW:
Groups:
- Cobomarsen (Randomized): Cobomarsen was administered by intravenous 2-hour infusion at a dose of 282 mg of the active moiety (equivalent to 300 mg of the active pharmaceutical ingredient or sodium salt form) on Days 1, 3, 5, 8, and weekly thereafter. Cobormarsen: 282 mg 2 hour IV infusion
- Vorinostat (Randomized): Vorinostat (400 mg [4x100 mg capsules]) was administered orally once daily with food, at approximately the same time each day. Subjects with abnormal alanine aminotransferase/ aspartate aminotransferase (ALT/AST) (> upper limit of normal [ULN]) or bilirubin (> 1.0 × ULN) at screening were to start vorinostat dosing at 300 mg (three 100-mg capsules) once daily with food, at approximately the same time each day, per dosing guidelines.
  Vorinostat: 100 mg capsules
- Cobomarsen (Crossover): For subjects that were randomized to Vorinostat during the randomized period and were eligible to receive Cobomarsen during the crossover period: Cobomarsen was administered by intravenous 2-hour infusion at a dose of 282 mg of the active moiety (equivalent to 300 mg of the active pharmaceutical ingredient or sodium salt form) on Days 1, 3, 5, 8, and weekly thereafter. Cobormarsen: 282 mg 2 hour IV infusion
Period: Randomized Period
Arm/Group | Cobomarsen (Randomized) | Vorinostat (Randomized) | Cobomarsen (Crossover)
Started | 19 | 18 | 0
Completed | 4 | 8 | 0
Not Completed | 15 | 10 | 0
Not completed — Adverse Event | 1 | 5 | 0
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0
Not completed — Participant decision | 3 | 1 | 0
Not completed — Study terminated by sponsor | 6 | 3 | 0
Period: Cobomarsen Crossover Period
Arm/Group | Cobomarsen (Randomized) | Vorinostat (Randomized) | Cobomarsen (Crossover)
Started | 0 | 0 | 7
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 7
Not completed — Physician Decision | 0 | 0 | 2
Not completed — Sponsor Decision to terminate trial | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cobomarsen | Vorinostat | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 27
  >=65 years | 6 | 4 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 10 | 11 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 14 | 14 | 28
  Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 17 | 13 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 0 | 1
  Belgium | 2 | 3 | 5
  United States | 9 | 8 | 17
  Italy | 0 | 1 | 1
  United Kingdom | 4 | 2 | 6
  France | 1 | 3 | 4
  Spain | 2 | 1 | 3
Skin tumor at screening [Count of Participants; unit: Participants] | 6 | 4 | 10
No skin tumor at screening [Count of Participants; unit: Participants] | 13 | 14 | 27
Lactate dehydrogenase (LDH) is greater than upper limit normal (ULN) at diagnosis [Count of Participants; unit: Participants] | 4 | 2 | 6
LDH is not greater than ULN at diagnosis [Count of Participants; unit: Participants] | 15 | 14 | 29
LDH not reported at diagnosis [Count of Participants; unit: Participants] | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving an Objective Skin Response of at Least 4 Months Duration (ORR4)
Description: ORR4 is the percentage of subjects with a complete response (CR) or partial response (PR) in the skin for 4 consecutive months confirmed by repeat assessments no less than 28 days (± 3 days) later. The modified Severity Weighted Assessment Tool (mSWAT) is used to measure skin disease severity based on the percentage of body surface area (BSA) with patches, plaques, or tumors. Total scores are calculated by multiplying the BSA percentage for each category of lesion (patch, plaque, or tumor) by a weighting factor and adding the three sub-scores. Lower scores indicate a lower degree of skin disease severity. CR corresponds to 100% clearance of skin lesions present at baseline (mSWAT score of 0). PR corresponds to 50-99% clearance of skin disease present at baseline (at least 50% reduction in mSWAT score), without new tumors.
Time Frame: Date of first dose through the earlier of last study visit or interim analysis data cut-off date of 12-Oct-2020, up to 16 months
Population: Intent to treat population (includes all randomized subjects who received at least one dose of study treatment (cobomarsen or vorinostat) and had at least one post-baseline assessment. Assignment of subjects to treatment group is based on the planned treatment assignment.
Measure: Number; unit: Percentage of participants
Arm/Group | Cobomarsen (Randomized) | Vorinostat (Randomized)
Number analyzed (Participants) | 19 | 18
Percentage of participants | 15.8 | 16.7
Statistical Analysis 1: Comparison: Cobomarsen (Randomized) vs Vorinostat (Randomized); Comparison of the treatment groups is based on a Cochran-Mantel-Haenzel test controlling for the number of tumors at screening (at least one tumor at screening versus no tumors at screening) and number of prognostic factors (0-1 versus 2 prognostic factors). Prognostic factors include age at diagnosis > 60 years and lactate dehydrogenase level > upper limit of normal at diagnosis. Number of subjects achieving ORR4 and exact binomial (Clopper-Pearson) confidence intervals are presented; Test type: Superiority; p = .9539, Cochran-Mantel-Haenszel

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Time from date of randomization until the date of earliest documented progression or death from any cause. The duration of PFS was censored at the date of the last mSWAT assessment if the subject was alive and had no documented progression. Disease progression in the skin is defined as ≥ 25% increase in mSWAT score from baseline or, in participants with complete or partial response, increase in mSWAT score of greater than the sum of the nadir plus 50% baseline score.
Time Frame: Date of first dose through interim analysis data cut-off date of 12-Oct-2020, up to 16 months
Population: Intent to treat population (includes all randomized subjects who received at least one dose of study treatment [cobomarsen or vorinostat] and had at least one post-baseline assessment). Assignment of subjects to treatment group is based on the planned treatment assignment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cobomarsen (Randomized) | Vorinostat (Randomized)
Number analyzed (Participants) | 19 | 18
months | NA [9.26 to NA] — Median is defined to be the smallest observed survival time for which the value of the estimated survival function is less than or equal to 0.5. The median could not be calculated from the available data because there were an insufficient number of participants with events. | 6.01 [2.89 to 8.90]
Statistical Analysis 1: Comparison: Cobomarsen (Randomized) vs Vorinostat (Randomized); Hazard ratio (cobomarsen/vorinostat) and p-value comparing the treatment groups is based on a Cox proportional hazards model. A hazard ratio < 1 favors cobomarsen over vorinostat; Test type: Superiority; p = 0.011, Regression, Cox

3. Secondary Outcome: Complete Response Rate
Description: Percentage of subjects with a complete response in the skin based on mSWAT
Time Frame: Date of first dose through interim analysis data cut-off date of 12-Oct-2020, up to 16 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Cobomarsen (Randomized) | Vorinostat (Randomized)
Number analyzed (Participants) | 19 | 18
Percentage of participants | 0 | 5.6

4. Secondary Outcome: Time to Progression
Description: Time from date of randomization until the earliest date of confirmed progression
Time Frame: Date of first dose through interim analysis data cut-off date of 12-Oct-2020, up to 16 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Cobomarsen (Randomized) | Vorinostat (Randomized)
Number analyzed (Participants) | 19 | 18
Months | NA [9.26 to NA] — Median could not be calculated from the available data. | 6.01 [2.89 to 8.90]

5. Secondary Outcome: Time to Maximal Effect in mSWAT
Description: Time to greatest improvement in mSWAT score
Time Frame: Monthly from first dose through interim analysis data cut-off date of 12-Oct-2020, up to 16 months
Population: Participants with improvement in mSWAT score
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Cobomarsen (Randomized) | Vorinostat (Randomized)
Number analyzed (Participants) | 17 | 14
Months | 4.5 (3.7) | 3.0 (2.7)

6. Secondary Outcome: Objective Response Rate in the Skin of at Least 28-days Duration (ORR1)
Description: Percentage of participants achieving ≥ 50% improvement in mSWAT of at least 28-days duration
Time Frame: Monthly from first dose through interim analysis data cut-off date of 12-Oct-2020, up to 16 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Cobomarsen (Randomized) | Vorinostat (Randomized)
Number analyzed (Participants) | 19 | 18
percentage of participants | 31.6 | 33.3

7. Secondary Outcome: Percentage of Subjects Achieving ≥ 50% Improvement in mSWAT at 28 Days
Description: Percentage of subjects achieving ≥ 50% improvement from baseline in mSWAT at 28 days after first dose
Time Frame: 28 days after first dose
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Cobomarsen (Randomized) | Vorinostat (Randomized)
Number analyzed (Participants) | 19 | 18
percentage of participants | 5.3 | 11.1

8. Secondary Outcome: Percentage of Subjects Achieving ≥ 50% Improvement in mSWAT at 4 Months
Description: Percentage of subjects achieving ≥ 50% improvement from baseline in mSWAT at 4 months after first dose
Time Frame: 4 months after first dose
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Cobomarsen (Randomized) | Vorinostat (Randomized)
Number analyzed (Participants) | 19 | 18
percentage of participants | 21.1 | 22.2

9. Secondary Outcome: Time to ≥ 50% Improvement in mSWAT
Description: Time from date of randomization until ≥ 50% improvement in mSWAT score
Time Frame: Monthly from first dose through interim analysis data cut-off date of 12-Oct-2020, up to 16 months
Population: Subjects who achieved an objective response in skin (≥ 50% improvement in mSWAT)
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Cobomarsen (Randomized) | Vorinostat (Randomized)
Number analyzed (Participants) | 6 | 6
Months | 3.7 (2.7) | 2.7 (1.8)

10. Secondary Outcome: Duration of Response in Skin
Description: Duration of response in skin (no progression after achieving ≥ 50% improvement in mSWAT)
Time Frame: Monthly from first dose through interim analysis data cut-off date of 12-Oct-2020, up to 16 months
Population: Subjects who achieved an objective response in skin (≥ 50% improvement in mSWAT)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cobomarsen (Randomized) | Vorinostat (Randomized)
Number analyzed (Participants) | 6 | 6
Months | NA [NA to NA] — Median was defined as the smallest observed survival time for which the value of the Kaplan-Meier estimated survival function was less than or equal to 0.5. The median and 95% Confidence Interval could not be calculated from the available data. | 7.85 [6.60 to NA] — Median was defined as the smallest observed survival time for which the value of the Kaplan-Meier estimated survival function was less than or equal to 0.5. The 95% Confidence Interval could not be calculated from the available data.

11. Secondary Outcome: Pruritus Medication Utilization
Description: Change from baseline in number of pruritus medications taken per subject
Time Frame: Date of first dose through end of treatment or interim analysis data cut-off date of 12-Oct-2020, up to 16 months
Population: All subjects with any predose or postdose pruritus medications, including subjects with no predose medications and at least one postdose medication
Measure: Mean (Standard Deviation); unit: Number of pruritus medications
Arm/Group | Cobomarsen (Randomized) | Vorinostat (Randomized)
Number analyzed (Participants) | 14 | 7
Number of pruritus medications | -1 (2.39) | -0.9 (1.35)

12. Other Pre Specified Outcome: Peak Plasma Concentration (Cmax) of Cobomarsen - First Dose
Description: Peak plasma concentration (Cmax) of cobomarsen after first dose
Time Frame: 1, 1.92, 6, 24 and 48 hours post-dose after the first dose
Population: Population analyzed included those randomized to cobomarsen treatment.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Cobomarsen (Randomized)
Number analyzed (Participants) | 19
µg/mL | 10.5 (7.17)

13. Other Pre Specified Outcome: Peak Plasma Concentration (Cmax) of Cobomarsen - Week 5
Description: Peak plasma concentration (Cmax) of cobomarsen after fourth dose (Week 5)
Time Frame: 1, 1.92 and 6 hours post-dose after the Week 5 dose
Population: Population analyzed included those randomized to cobomarsen treatment.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Cobomarsen (Randomized)
Number analyzed (Participants) | 19
µg/mL | 9.34 (3.24)

14. Other Pre Specified Outcome: Area Under the Plasma Concentration vs. Time Curve (AUC) of Cobomarsen - Week 5
Description: Area under the curve (AUClast) for cobomarsen plasma concentration versus time curve after the fourth (Week 5) dose
Time Frame: 1, 1.92 and 6 hours post-dose after the Week 5 dose
Population: Population analyzed included those randomized to cobomarsen treatment.
Measure: Mean (Standard Deviation); unit: µg*hr/mL
Arm/Group | Cobomarsen (Randomized)
Number analyzed (Participants) | 19
µg*hr/mL | 25.5 (6.27)

15. Other Pre Specified Outcome: Number of Participants With Anti-drug Antibody Generation
Description: Number of participants who develop antibodies to cobomarsen during treatment
Time Frame: Date of first dose through interim analysis data cut-off date of 12-Oct-2020, up to 16 months
Population: The study was prematurely terminated for business reasons. No data were collected to evaluate this endpoint.
Arm/Group | Cobomarsen (Randomized) | Vorinostat (Randomized)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) that occurred from the time of informed consent through the last study visit, up to 18 months
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research. Treatment emergent AEs (those occurring after the first dose of study medication) are reported.
Groups:
- Cobomarsen (Randomized): Cobomarsen was administered by intravenous 2-hour infusion at a dose of 282 mg of the active moiety (equivalent to 300 mg of the active pharmaceutical ingredient or sodium salt form) on Days 1, 3, 5, 8, and weekly thereafter. Cobomarsen: 282 mg 2 hour IV infusion
- Cobomarsen (Crossover): For subjects that were randomized to Vorinostat during the randomized period and were eligible to receive Cobomarsen during the crossover period: Cobomarsen was administered by intravenous 2-hour infusion at a dose of 282 mg of the active moiety (equivalent to 300 mg of the active pharmaceutical ingredient or sodium salt form) on Days 1, 3, 5, 8, and weekly thereafter. Cobomarsen: 282 mg 2 hour IV infusion
Arm/Group | Cobomarsen (Randomized) | Vorinostat (Randomized) | Cobomarsen (Crossover)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18 | 0/7
Serious Adverse Events (participants affected / at risk) | 2/19 | 1/18 | 0/7
Other Adverse Events (participants affected / at risk) | 18/19 | 18/18 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cobomarsen (Randomized) (N=19) | Vorinostat (Randomized) (N=18) | Cobomarsen (Crossover) (N=7)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Superinfection of Skin Lesions (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cobomarsen (Randomized) (N=19) | Vorinostat (Randomized) (N=18) | Cobomarsen (Crossover) (N=7)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (2) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (6) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Bacterial test positive (Investigations) | 1 (2) | 0 (0) | 0 (0)
Blood alkaline phosphatase increase (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (4) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Blood pressure decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 2 (3) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (3) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Crystal urine present (Investigations) | 0 (0) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 7 (9) | 8 (10) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (5) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 0 (0)
Ear infection (Infections and infestations) | 1 (3) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 1 (3) | 0 (0) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 7 (12) | 6 (10) | 2 (2)
Feeling cold (General disorders) | 1 (1) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastoenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 5 (7) | 1 (1) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (10) | 5 (15) | 2 (3)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (Infections and infestations) | 2 (2) | 3 (4) | 0 (0)
Infusion site pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (7) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (10) | 6 (7) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Overgrowth bacterial (Infections and infestations) | 2 (3) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extermity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0)
Parosmia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (20) | 4 (4) | 0 (0)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus generalized (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Red blood cells urine positive (Investigations) | 1 (1) | 1 (2) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Skin bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (7) | 1 (1) | 0 (0)
Skin infection (Skin and subcutaneous tissue disorders) | 5 (18) | 0 (0) | 0 (0)
Skin plaque (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin weeping (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Superinfection (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Superinfection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (4)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (4) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3) | 0 (0)
Tumour inflammation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Urine abnormality (Renal and urinary disorders) | 1 (2) | 1 (1) | 0 (0)
Urine albumin/creatinine ratio increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early for business reasons, and not due to concerns regarding safety or lack of efficacy. Because the study was terminated early, enrollment was ended at 37 participants instead of the initially planned 126 participants, and a planned interim analysis based on these 37 participants was the only analysis performed for the study. The study duration was also shortened from an estimated 36 months to 20 months overall.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators in this study may present or publish study results in scientific journals or other scholarly media without prior written approval after the following conditions have been met:

* Results of study have been publicly disclosed by or with the consent of the sponsor
* Investigator has complied with the Clinical Trial Agreement and requests from the sponsor to delete confidential information (other than study results)
* Study has been completed at all study sites for at least 2 years

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-10): https://cdn.clinicaltrials.gov/large-docs/20/NCT03713320/Prot_SAP_000.pdf